CLINICAL TRIAL: NCT00535613
Title: Does a Single Dose of Propofol Decrease the Incidence of Emergence Agitation in Children?
Brief Title: Propofol in Emergence Agitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2007-0069
Record Dates: First submitted 2007-09-23; First posted 2007-09-26 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): propofol
  Interventions: Drug: Propofol
- 2 (Sham Comparator): no propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — IV, single bolus at completion of anesthetic, 0.1 ml/kg

SUMMARY:
The purpose of the study is to see if a small dose of propofol given intravenously (through a needle into a vein) at the end of anesthesia can make it less likely that children will be agitated as the come out of the anesthetic.

DETAILED DESCRIPTION:
Emergence agitation is defined as a mental disturbance during the recovery from general anesthesia. It consists of confusion, disorientation, delusions, and hallucinations. It manifests in children as some combination of restlessness, moaning, inconsolable crying, involuntary physical activity, and thrashing about. This puts patients at risk of injuring themselves or their caregivers, causing bleeding or disruption of their surgical repair, and pulling out IVs and drains. It can be difficult to maintain necessary vital sign monitoring in these agitated patients, and constant one-on-one nursing is often required. When emergence agitation occurs, all members of the healthcare team, and the parents report dissatisfaction with the quality of the child's recovery from anesthesia.

Propofol is a commonly used intravenous anesthetic agent. Studies have compared continuous infusions of intravenous propofol versus inhalational sevoflurane for the maintenance of anesthesia. These have shown a significant decrease in the incidence of emergence agitation in the patients who received the propofol infusions. This proposed study will investigate the effects of a single bolus dose of propofol at the conclusion of a sevoflurane inhalational anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12 months to 6 years old
* Planned surgery/procedure: The goal is to enroll patients who will not have pain when they awake from anesthesia. We will include patients who are having magnetic resonance imaging (MRI) under anesthesia, or an eye exam under anesthesia. We will also include those patients who are having a surgery in which a regional or caudal block is part of the planned anesthetic. This will be small orthopedic procedures in the lower extremities; or urologic or general surgical procedures below the level of the umbilicus. These patients have been chosen because the regional/caudal block should result in the patient not having pain when they awake from anesthesia.

(The caudal block is a single epidural injection of local anesthetic that is done when the pediatric patient is under general anesthesia. It is a routine procedure that results in numbness below the level of the umbilicus, and gives relief of pain, for about 8 hours.)

Examples of orthopedic surgeries include, but are not limited to:

Removal of an extra digit or syndactyly repair Club foot releases Lower extremity tendon releases or lengthenings Lower extremity tendon transfers Removal of hardware

Examples of urologic surgeries include, but are not limited to:

Circumcision or circumcision revision hypospadias repair Chordee repair Orchiopexy Orchiectomy

Examples of general pediatric surgeries include, but are not limited to:

Inguinal hernia repair Rectal muscle biopsies Excision of lower extremity or lower abdominal mass Burn scar releases and skin grafting

Exclusion Criteria:

* Obstructive sleep apnea-Patients with sleep apnea are not ideal candidates for removal of their endotracheal tube or laryngeal mask airway while still somewhat anesthetized. It is preferable to extubate these patients awake.
* Developmental delays-Patients with developmental delays may not interact with their environment, make eye contact, have purposeful actions, or be aware of their surroundings even when at their baseline pre-operatively. It would be difficult to evaluate these features of emergence agitation in children who demonstrate this behavior on a routine basis.
* Psychological disorders-Patients with psychological disorders may have the same issues as those with developmental delays when it comes to evaluating their behavior after anesthesia.
* Egg white allergy-Propofol is contraindicated in patients with egg white allergies due to risk of allergy to the propofol lecithin base.

Ages: 12 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cari Meyer, MD, Principal Investigator — Univeristy of Wisconsin - Madison
Locations (1):
- Univeristy of Wisconsin - Madison, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: No propofol
Period: Overall Study
Arm/Group | Propofol | Placebo
Started | 49 | 50
Completed | 49 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Placebo | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Mean (Full Range); unit: years] | 1.88 [1 to 5] | 1.72 [1 to 6] | 1.80 [1 to 6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 47 | 48 | 95
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Emergent Agitation
Description: Incidence of Emergent Agitation is defined as a Paediatric Anaesthesia Emergence Delirium (PAED) score above 10 at any point at the defined protocol time points (recovery, 5, 10, 15, 20, 25, or 30 minutes)
Time Frame: up to 30 min post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol | Placebo
Number analyzed (Participants) | 49 | 50
Participants | 16 | 24

2. Secondary Outcome: Time Spent in Recovery Room
Time Frame: up to 1 hour post surgery
Population: The study team planned to collect post anesthesia care unit discharge time from the subject medical records, however PACU discharge time was often not recorded in routine cases during the study period. This was not anticipated by the study team and retrospective analysis was not possible for this outcome.
Arm/Group | Propofol | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants Who Received Medication in the Recovery Room
Time Frame: up to 1 hour post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol | Placebo
Number analyzed (Participants) | 49 | 50
Participants | 3 | 6

ADVERSE EVENTS:
Time Frame: Up to 30 min post surgery
Arm/Group | Propofol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes